CLINICAL TRIAL: NCT03821233
Title: A Phase 1 Study of ZW49 in Patients With Locally Advanced (Unresectable) or Metastatic HER2-Expressing Cancers
Brief Title: A Dose Finding Study of ZW49 in Patients With HER2-Positive Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zymeworks BC Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZWI-ZW49-101
Record Dates: First submitted 2019-01-28; First posted 2019-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: HER2-expressing Cancers
Keywords: HER2; Bispecific antibody; Biparatopic antibody; Immunotherapy; Gastric cancers; Esophageal cancers; Gastroesophageal junction (GEJ) cancers; Breast cancer; Ovarian cancer; Non-small cell lung cancer; Colorectal cancer; Cholangiocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZW49 (Experimental)
  Interventions: Drug: ZW49

INTERVENTIONS:
Drug: ZW49 — * Dose Escalation: ZW49 administered intravenously at dose levels determined by the SMC
  * Expansion: MTD or RD identified in the dose-escalation part of the study

SUMMARY:
This is a first-in-human, Phase 1, multicenter, open-label, dose-escalation study to establish the maximum-tolerated dose (MTD) or recommended dosage (RD) of ZW49, the investigational agent under study, and to assess the safety and tolerability of ZW49. Eligible patients include those with locally advanced (unresectable) or metastatic HER2-expressing cancers.

DETAILED DESCRIPTION:
The study will use a 3+3 dose-escalation study design to evaluate the safety and tolerability of ZW49 and to determine the MTD or RD of ZW49 for further study. Selected expansion cohorts will be subsequently opened based upon Safety Monitoring Committee (SMC) recommendation and sponsor approval to further evaluate the safety and tolerability of ZW49 at the MTD or RD and to assess preliminary anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-confirmed diagnosis of breast cancer, gastroesophageal adenocarcinoma (GEA), or other HER2-expressing cancer with evidence of locally advanced (unresectable) and/or metastatic disease.

  * Dose-escalation (Cohort 1): HER2-high advanced solid tumors
  * Expansion (Cohort 2): HER2-high breast cancer
  * Expansion (Cohort 3): HER2-high GEA
  * Expansion (Cohort 4): HER2-high other non-breast and non-GEA cancers
* Progressive disease that has progressed on or been refractory to all standard of care. Patients who were intolerant to or ineligible for standard therapy may be eligible if the reasons are carefully documented and approval is provided by the sponsor medical monitor

  * Patients with HER2-high breast cancer must have received prior treatment with trastuzumab, pertuzumab, and ado-trastuzumab emtansine (T-DM1)
  * Patients with HER2-high GEA must have received prior treatment with trastuzumab
* Sites of disease assessible per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

  * Dose-escalation: measurable or non-measurable disease
  * Expansion: measurable disease
* ECOG performance status score of 0 or 1
* Adequate organ function
* Adequate cardiac left ventricular function, as defined by a LVEF >/= institutional standard of normal

Exclusion Criteria:

* History of myocardial infarction or unstable angina within 6 months prior to enrollment, troponin levels consistent with myocardial infarction, or clinically significant cardiac disease, such as ventricular arrhythmia requiring therapy, uncontrolled hypertension, or any history of symptomatic congestive heart failure (CHF)
* Clinically significant infiltrative pulmonary disease not related to lung metastases
* Active hepatitis B or hepatitis C infection or other known chronic liver disease
* Acute or chronic uncontrolled renal disease, pancreatitis, or liver disease (with exception of patients with Gilbert's Syndrome, asymptomatic gall stones, liver metastases, or stable chronic liver disease per investigator assessment)
* Known history of human immunodeficiency virus (HIV) infection
* Brain metastases: Untreated CNS metastases, symptomatic CNS metastases, or radiation treatment for CNS metastases within 4 weeks of start of study treatment. Stable, treated brain metastases are allowed (defined as patients who are off steroids and anticonvulsants and are stable for at least 1 month at the time of screening).
* Known leptomeningeal disease (LMD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | Up to 4 weeks
  Number of participants who experienced a DLT. DLTs are events that occur following administration of any amount of ZW49 and are considered related to ZW49 per the investigator. DLTs will include only events considered related to ZW49.
Incidence of adverse events | Up to 7 months
  Number of participants who experienced an adverse event
Incidence of lab abnormalities | Up to 7 months
  Number of participants who experienced a maximum severity of Grade 3 or higher post-baseline laboratory abnormality, including either hematology and chemistry. Grades are defined using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Incidence of electrocardiogram (ECG) and left ventricular ejection fraction (LVEF) abnormalities | Up to 7 months
  Number of participants who experienced an abnormal ECG or LVEF
Incidence of dose reductions of ZW49 | Up to 7 months
  Number of doses reduced and number of participants who require a dose reduction

SECONDARY OUTCOMES:
Serum concentrations of ZW49 | Up to 7 months
  End of infusion concentration, maximum serum concentration, and trough concentration of ZW49
Incidence of anti-drug antibodies (ADAs) | Up to 7 months
  Number of participants who develop ADAs
Objective response rate (ORR) | Up to 6 months
  Number of participants who achieved a best response of either complete or partial response during treatment according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Disease control rate | Up to 6 months
  Number of participants who achieved a best response of complete response, partial response, or stable disease during treatment according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Duration of response | Up to 2 years
  Median duration of response (in months) and range (minimum, maximum)
Progression-free survival | Up to 2 years
  Median progression-free survival (in months) and range (minimum, maximum)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Woolery, PharmD, BCOP, Study Director — Zymeworks BC Inc.
Locations (16):
- United States (8):
  - City of Hope, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Flinders Medical Centre, Adelaide, Australia
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No